CLINICAL TRIAL: NCT02863757
Title: Disease Progression and Clinical Outcomes in Chronic Hepatitis B (CHB) Patients With Comorbid Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: Follow-up of Chronic Hepatitis B Patients With Comorbid Nonalcoholic Fatty Liver Disease
Status: Recruiting | Type: Observational
Sponsor: Humanity and Health Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: H&H_NAFLD/CHB
Record Dates: First submitted 2016-08-04; First posted 2016-08-11 (Estimated); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chronic Hepatitis B; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Hepatitis B, Chronic; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- CHB Group: Patients with chronic hepatitis B
- CHB/NAFLD Group: Patients with chronic hepatitis B and comorbid nonalcoholic fatty liver disease
- NAFLD Group: Patients with nonalcoholic fatty liver disease

SUMMARY:
The purpose of this study is to determine the disease progression in CHB/NAFLD compared with CHB and NAFLD including liver cirrhosis, cirrhotic complications and hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Liver biopsy proved CHB and/or NAFLD at baseline;
* Chinese
* Follow-up duration>12 months

Exclusion Criteria:

* Other liver diseases;
* Secondary causes of hepatic steatosis;
* Alcohol abuse;
* Liver cirrhosis, cirrhosis related complications or HCC at baseline;
* Malignancy;
* History of liver transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hosptials and primary care clinics
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with liver cirrhosis, hepatic encephalopathy, esophageal varices, ascites and hepatocellular carcinoma | Up to 20 years

SECONDARY OUTCOMES:
Number of patients with hypertension, obesity, diabetes mellitus, hyperlipidaemia | Up to 20 years
Number of patients with liver transplantation and liver-related death | Up to 20 years
Diagnosis time of liver cirrhosis, hepatic encephalopathy, esophageal varices, ascites and hepatocellular carcinoma from baseline | Up to 20 years
Occurrence time of liver transplantation and liver-related death from baseline | Up to 20 years

CONTACTS AND LOCATIONS:
Locations (1):
- Humanity and Health GI and Liver Centre, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No